CLINICAL TRIAL: NCT00717015
Title: Tamoxifen Pharmacokinetics and CYP2D6 Polymorphisms in Asian Women With Hormone Receptor Positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR02/06/06
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Hormone Receptor Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
We hypothesized that subjects with CYP2D6*10 alleles may have a lower steady state levels of endoxifen due to reduced conversion of tamoxifen to endoxifen.

Primary objectives:

* To determine the steady state pharmacokinetics of tamoxifen and its metabolites
* To test the effects of genetic polymorphisms of CYP2D6 on plasma concentration of tamoxifen and its metabolites in hormone receptor positive women who are taking tamoxifen as adjuvant treatment for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* At least 18 years of age.
* On tamoxifen for at least 3 months for adjuvant therapy.
* On a stable diet for past 1 week before blood sampling.
* Compliant with tamoxifen medication.
* Completed adjuvant chemotherapy and/or adjuvant radiation therapy.

Exclusion Criteria:

• Patients should not be on the list of medications for the last 1 week before accrual to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to enroll 200 patients onto our study over a period of 2 years. Patients will be recruited from the oncology outpatient clinic in National University Hospital. Participation in the study will be strictly voluntary and written informed consent will be obtained from all subjects according to institutional and governmental guidelines. Consent will be obtained by attending doctors or co-investigators of the study prior to blood sampling.
Sampling Method: Probability Sample
Dates: Start 2005-11

PRIMARY OUTCOMES:
To determine the steady state pharmacokinetics of tamoxifen and its metabolites
To test the effects of genetic polymorphisms of CYP2D6 on plasma concentration of tamoxifen and its metabolites in hormone receptor positive women who are taking tamoxifen as adjuvant treatment for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Chiung Ing Wong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore